CLINICAL TRIAL: NCT03285581
Title: Open-label, Prospective, Multicenter Pivotal Study of the Cutera truSculpt™ Radiofrequency Device for Wrinkle Reduction
Brief Title: Pivotal Study of the Cutera truSculpt Radiofrequency Device for Wrinkle Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-17-TS14
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Wrinkle Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- truSculpt RF (Other): Subjects will receive RF treatments
  Interventions: Device: truSculpt RF

INTERVENTIONS:
Device: truSculpt RF — Subjects will receive RF treatments
  Other Names: Device: Treatment

SUMMARY:
The purpose of this pivotal investigation is to evaluate the safety and efficacy of the Cutera truSculpt™ radiofrequency (RF) Device for Wrinkle Reduction.

DETAILED DESCRIPTION:
This is an Open-label, Prospective, Multicenter Pivotal Study of approximately 40 male or female subjects, age 25 to 65 years who desire RF treatment for wrinkle reduction and improvement in skin quality. Subjects will receive RF treatments with the Cutera truSculpt™ radiofrequency (RF) device. Subjects will return to the site after study treatments have been delivered 12 weeks post-final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and provide written informed consent and release of health information
2. Male or Female, 25 to 65 years of age (inclusive)
3. Fitzpatrick Skin Type I - VI (Appendix 4)
4. Has visible wrinkles or skin laxity in the treatment area
5. On the Fitzpatrick Classification Wrinkle Classification System subject has a pre-treatment score of 4-9 (inclusive) (Appendix 5)
6. No use of tobacco products for at least 6 months and willing to refrain from use for the duration of the study
7. Subject must agree to not undergo any other cosmetic procedure(s) area, or start topical retinol products in the treatment area during the study period
8. Subject must be willing to adhere to the follow-up schedule and study instructions
9. Subject must be willing to adhere to the same diet and/or exercise routine throughout the study, and agree to maintain the same weight throughout the study, within 10% of baseline weight measurement
10. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentations, educational, and/or marketing purposes
11. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant -

Exclusion Criteria:

1. Participation in a clinical trial of a drug or another device in the target area within 3 months of study participation, or during the study.
2. Any type of prior cosmetic treatment to the target area within 12 months of study participation e.g., radiofrequency, cryolipolysis, deoxycholate injection, or light-based treatments
3. Prior injection of botulinum toxin, collagen, hyaluronic acid filler, or other dermal filler, and medium-depth to deep chemical peels, to the treatment area within 6 months of study participation
4. History of systemic steroid use within 3 months; history of topical steroid use in the target area within 2 months
5. History of systemic retinoid (isotretinoin) and therapeutic dose of Vitamin A within 6 months of study participation
6. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant
7. Has metal implant(s) within the body that are local to the treatment area, such as surgical clips, plates and screws (metal tooth fillings or crowns will not exclude subject participation), or has , artificial heart valves or artificial joints
8. Clinically significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders that in the opinion of the Investigator will confound participation in the study
9. Diagnosed or documented immune system disorders
10. History of any disease or condition that could impair wound healing
11. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen
12. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing
13. Infection, dermatitis, rash or other skin abnormality in the target area
14. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation
15. Anticipated or planned need for surgery or hospitalization during the duration of the study
16. Pregnant, nursing, or planning a pregnancy during the trial; or is a woman of child bearing potential but is not willing to use an acceptable method of contraception as determined by the Investigator
17. As per the Investigator's discretion, any physical or psychological condition which might make it unsafe for the subject to participate in this study -

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, M.D., Principal Investigator — Cutera Research Center; Daniel Friedmann, M.D., Principal Investigator — Westlake Dermatology
Locations (2):
- United States (2):
  - Cutera Research Center, Brisbane, California
  - Westlake Dermatology, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm-1: Subject(s) will receive RF treatments
Period: Overall Study
Arm/Group | Arm-1
Started | 39
Completed | 25
Not Completed | 14

BASELINE CHARACTERISTICS:
Groups:
- truSculpt RF: Subject will receive RF treatments
Arm/Group | truSculpt RF
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Principal Investigator's Assessment of Improvement at 12 Weeks Post-final Treatment (Physician's Global Assessment of Improvement=GAIS)
Description: GAIS: 4=Very Significant Improvement, 3=Significant Improvement, 2=Moderate Improvement, 1=Mild Improvement, 0=No Change Higher scores indicate better outcomes
Time Frame: 12 weeks post-final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | truSculpt RF
Number analyzed (Participants) | 25
score on a scale | 1.04 (0.45)

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment, up to 7 months
Arm/Group | truSculpt RF
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 39/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | truSculpt RF (N=39)
Erythema (Skin and subcutaneous tissue disorders) | 39
Edema (Skin and subcutaneous tissue disorders) | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03285581/Prot_SAP_000.pdf